CLINICAL TRIAL: NCT07171489
Title: An Early Feasibility Study of Using the AccelBand, a Leg-worn Transcutaneous Neuromodulation (TNM) Device, for Neurogenic Bowel Dysfunction (NBD) in People With Spinal Cord Injury (SCI)
Brief Title: Efficacy of a Wearable Noninvasive Neuromodulation Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gianna Rodriguez, Clinical Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00279126; 1UG3NS125182-01 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
Keywords: Neurogenic bowel dysfunction; Transcutaneous neuromodulation; Questionnaires; AccelBand; Anorectal manometry test
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomized 4-week treatment period will be double-blinded for TNM and sham-TNM except for the study coordinator. Participants are unblinded at the 4-week post treatment visit. Of note, sham participants have the option of having a 2-week open label of treatment following the randomized treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham (TNM at a sham-point) -Randomized arm (Sham Comparator): Participants will have a 2-week phase-in period.followed by a 4-week sham treatment.
  Sham participants can elect to have 2 weeks of open-label treatment once unblinded after 4 weeks of sham.
  Interventions: Device: TNM at a sham-point (AccelBand) - randomized arm; Device: TNM at a leg point (AccelBand)- open-label
- Transcutaneous neuromodulation (TNM) at a leg point-Randomized arm (Experimental): Participants will have a 2-week phase-in period followed by a 4-week treatment phase.
  Interventions: Device: TNM at a leg point (AccelBand)- randomized arm

INTERVENTIONS:
Device: TNM at a sham-point (AccelBand) - randomized arm — This will be self-administrated by study participants (or caregivers) for a period of approximately 4 weeks twice a day (once in the morning and once in the evening daily), each lasting 60 minutes. Scheduled weekly phone calls will be provided by the study team member to assure compliance with the TNM administration and answer any questions that a participant may have.
  In addition to the treatment period participants will have tests completed (baseline and following treatment), as well as complete surveys during the trial.
  Arms: Sham (TNM at a sham-point) -Randomized arm
Device: TNM at a leg point (AccelBand)- randomized arm — This will be self-administrated by study participants (or caregivers) for a period of approximately 4 weeks twice a day (once in the morning and once in the evening daily), each lasting 60 minutes. Scheduled weekly phone calls will be provided by the study team member to assure compliance with the TNM administration and answer any questions that a participant may have.
  In addition to the treatment period participants will have tests completed (baseline and following treatment), as well as complete surveys during the trial.
  Arms: Transcutaneous neuromodulation (TNM) at a leg point-Randomized arm
Device: TNM at a leg point (AccelBand)- open-label — After 4 weeks of blinded treatment sham participants will be given the option to continue open-label TNM treatment at a leg point acupoint. Participants that agree to this will be re-trained and allowed to keep the AccelBand for another 2 weeks. During this stage, participants will be asked to complete daily home-based TNM treatment and complete the daily online symptom questionnaires. Participants will complete a visit following this additional treatment.
  Arms: Sham (TNM at a sham-point) -Randomized arm

SUMMARY:
The aim of this study is to investigate the potential of transcutaneous neuromodulation (TNM) to treat slow colonic transit and constipation, termed the Neurogenic bowel dysfunction (NBD), in people with SCI. In this project, the study team will investigate the impact of an active treatment intervention vs. a sham control intervention on NBD symptoms in patients with SCI.

The study hypotheses:

* The proposed TNM treatment at a leg point will reduce NBD symptoms between baseline and post-therapy, when compared to the sham-TNM treatment.
* The therapeutic effect of TNM to improve the NBD symptoms is associated with improvement of the autonomic function in SCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic spinal cord injury (SCI)
* SCI level above the twelfth thoracic vertebra (T12)
* SCI classified as Sensory Incomplete (AIS B), C, or D
* Post-SCI time ≥ 6 months;
* Neurogenic bowel dysfunction (NBD) as a result of SCI
* Willing to sign the informed consent form

Exclusion Criteria:

* Significant cognitive impairment, impeding the ability to provide informed consent or complete the questionnaire
* Prior gastrointestinal surgeries other than uncomplicated appendectomies, cholecystectomy or cesarean sections
* Known diagnosis of diabetes mellitus
* Known current or past severe significant psychiatric disorder
* Known current substance abuse
* Implanted medical devices for electrical stimulation (e.g. cardiac pacemaker)
* Taking opioid medications on a regular daily basis
* Currently pregnant or actively planning a pregnancy
* Active inflammatory bowel disease
* Ventilator dependency
* Severe autonomic dysreflexia
* No preservation of the sacral spinal reflexes: bulbocavernosus, patella, or Achilles
* Complete absence of sensation in the leg (since it is needed for calibrating the TNM intensity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
The Neurogenic Bowel Dysfunction (NBD) score | Baseline (phase-in) to 4-week visit
  The scoring the degree of NBD symptoms and bowel routines, including frequency of bowel movements (0, 1 or 6 points), headache, perspiration or discomfort before or during defecation (0 or 2 points), medications for constipation (0, to 4 points), time used for each defecation (0, 3 or 7 points), frequency of digital stimulation or evacuation (0, 6 points), frequency of fecal incontinence (0, 6, 7 or13 points), medication for fecal incontinence (0, or 4 points), flatus incontinence (0 pr 2 points) and perianal skin problems (0 or 3 points). The score range is between 0-47 with a higher score meaning greater bowel dysfunction.
Prolonged colonic transit measurement to assess NBD severity | Baseline and approximately the 4-week post treatment visit
  This will be assessed using abdominal X-ray (which will allow researchers to evaluate participants bowel activity over time) as the retention of radiopaque markers after ingestion of one gelatin capsule with 24 radiopaque markers, 72 hours before visit.

SECONDARY OUTCOMES:
Daily Medication use for neurogenic bowel use | Baseline (phase-in) to 4-week visit
  Use of medications: name, dose, frequency of medications and duration.
Bowel routine techniques | Baseline (phase-in) to 4-week visit
  Duration and types of bowel routine techniques will be tracked by the bowel diary application (app).
Number of bowel movements per week | Baseline (phase-in) to 4-week visit
  This will be tracked by the bowel diary application (app).
Bristol stool form scale (BSFS) | Baseline (phase-in) to 4-week visit
  Bristol stool form scale scores the stool appearance for each bowel movement as proxy for colonic transit based on stool consistency (hard (1) to liquid (7) and shape tracked by the bowel diary app.
SCI Quality of Life Bowel Management Difficulties survey (SCI QoL-BMD) | Baseline (phase-in) to 4-week visit
  This survey has 26 questions with scoring of 15 factors related to feelings of distress associated with bowel management difficulties in the past week scored from 1 ("none at all" or "never") to 5 ("very much" or "always") to create the overall range of (26-130) with a higher score indicting lower quality of life.
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline (phase-in) to 4-week visit
  This scare uses a 7-point Likert type scale from 1 (no discomfort) to 7(very severe discomfort) to rate 15 symptom items including both upper and lower abdominal symptoms. There is a range of scores from 15-105 with a higher score indicating more discomfort.
Number of Adverse events (serious and non-serious) | Baseline to post treatment visit (approximately 4 weeks)
  The severity, relatedness, and expectedness will be noted (per protocol) by the following:
  * Mild, Moderate, Severe
  * Relationship to study products: Associated or Not associated
  * Expected or unexpected
Fecal loading in the colon | Baseline and approximately the 4-week post treatment visit
  This will be scored from 1 to 5 from the abdominal X-rays, where: 1 - none, 2 - mild, 3 - moderate, 4 - severe, and 5 - severe with colon dilatation.
Anorectal Manometry Test (AMT) - sensory thresholds | approximately 4-week post treatment visit
  This will be assessed at the clinic with anorectal manometry (ARM) during rectal balloon distention, sensory thresholds for the first sensation, urge to defecation, and maximal tolerance.
Anorectal Manometry Test (AMT) - rectal inhibitory reflex | approximately 4-week post treatment visit
  This will be assessed at the clinic with anorectal manometry (ARM).
Anorectal Manometry Test (AMT) - external anal sphincter (EAS) and rectum pressures at rest and during strain | approximately 4-week post treatment visit
  This will be assessed at the clinic with Anorectal manometry (ARM).
Anorectal Manometry Test (AMT) - Paradoxical external anal sphincter contraction | approximately 4-week post treatment visit
  This will be assessed at the clinic with Anorectal manometry (ARM).

CONTACTS AND LOCATIONS:
Overall Officials: Gianna Rodriguez, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No